CLINICAL TRIAL: NCT06693284
Title: A Window of Opportunity Trial of Mirdametinib Plus Vorinostat for NF1 Associated, H3K27 Trimethylation Deficient Malignant Peripheral Nerve Sheath Tumor [MPNST]
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022LS040
Record Dates: First submitted 2024-10-17; First posted 2024-11-18 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Primary Malignant Peripheral Nerve Sheath Tumors
MeSH Terms: interventions — mirdametinib; Vorinostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): newly diagnosed, PRC2 deficient, primary malignant peripheral nerve sheath tumors (MPNSTs)
  Interventions: Drug: mirdametinib and vorinostat

INTERVENTIONS:
Drug: mirdametinib and vorinostat — short course of the combination of mirdametinib and vorinostat prior to the most appropriate standard of care treatment for the patient's specific tumor (typically localized radiation followed by surgical resection).

SUMMARY:
This is a single center Phase 0 "window of opportunity" trial for the treatment of newly diagnosed, PRC2 deficient, primary malignant peripheral nerve sheath tumors (MPNSTs) with a short course of the combination of mirdametinib and vorinostat prior to the most appropriate standard of care treatment for their specific tumor (typically localized radiation followed by surgical resection). Four to eight patients, 12 years of age or older and meeting the study's biomarker inclusion criteria, would be enrolled onto this trial. After voluntary written consent (assent with parent consent for minors) the patient undergoes MRI and PET imaging of the tumor and a needle biopsy to collect tumor is performed. Patients with histone H3K27 trimethylation deficient MPNST, as confirmed by immunohistochemistry, receive a single 28-day course of mirdametinib and vorinostat at standard oral dosing for each. At day 26, 27, or 28 the patient returns to clinic for a research visit repeating the baseline MRI and PET imaging and the needle biopsy for tumor tissue.

This ends direct study participation. The patient goes on to the most appropriate standard of care treatment for their MPNST. Information about the subsequent standard of care treatment is collected for the purposes of this study.

ELIGIBILITY:
Inclusion Criteria:

* Known Neurofibromatosis type 1 (NF-1) syndrome based on current diagnostic criteria.
* Diagnosis of suspected MPNST by PET or MRI imaging
* Confirmation of histone H3 lysine 27 trimethylation-negative MPSNT by immunohistochemistry
* Twelve years of age or older
* Complete blood count (CBC), platelet, liver and kidney function within institutional normal limits performed within 14 days of 1 st dose of study drug.
* Must be able to swallow capsules.
* Females of childbearing potential must use highly effective contraception (see inclusion criteria section) from the time of study enrollment through 6 months after the last dose of vorinostat and mirdametinib. Males with partners of childbearing potential must use highly effective contraception from the time of study enrollment through 3 months after the last dose of vorinostat.
* Provides voluntary written consent prior to any study related activities, with parental/guardian consent and assent for those 12 to 17 years of age at enrollment.

Exclusion Criteria:

* Pregnant or breastfeeding - females of childbearing potential must have a negative pregnancy test (serum or urine) within 7 days prior to the 1 st dose of the study drugs.
* Significant cardiac disease
* Significant eye disease
* Radiation therapy or chemotherapy in the past year.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Assess the toxicity of the combination of mirdametinib and vorinostat in patients with NF1-associated high grade MPNSTs. | 48 months
  As a result of the vaccine, both unique CNS toxicity and edema have been previously observed as soon as 10 days from the initiation of therapy. Neurotoxicity ≤ Grade 3 is an expected risk of this treatment. This will be measured as the number of participants experiencing this adverse event.
Determine the response of therapeutic targets | 48 months
  measuring phospho-ERK and histone H3K27 acetylation in post-therapy tumor tissue as compared to pre-treatment tumor tissue.
Evaluate the utility of radiographic response to this regimen | 48 months
  using MRI and PET.
  Each patient will undergo MRI of the primary lesion and CT/PET scan for staging and assessment of FDG uptake in the tumor at diagnosis and after completing 28 days of therapy with mirdametinib and vorinostat. Each patient will have a diagnostic tumor biopsy performed as a condition of entry into the study and to measure specific molecular tumor markers. A second biopsy will be performed at the completion of protocol therapy to assess tumor response to the therapy and to see if the specific tumor markers have changed as a result of the therapy given.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Galvin, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States